CLINICAL TRIAL: NCT05017142
Title: Swiss Pediatric Inflammatory Bain Disease Cohort Study
Brief Title: Swiss Pediatric Inflammatory Brain Disease Registry (Swiss-Ped-IBrainD)
Status: Recruiting | Type: Observational
Sponsor: University of Bern (Other)
Collaborators: Schweizerische Multiple Sklerose Gesellschaft (Other); Insel Gruppe AG, University Hospital Bern (Other); Novartis (Industry); Anna Mueller Grocholski-Stiftung (Unknown); Gottfried und Julia Bangerter- Rhyner-Stiftung, Basel (Other); Biogen (Industry); Roche Pharma (Switzerland) Ltd (Unknown); Fondation Johanna Dürmüller-Bol (Unknown); Kantonsspital Aarau (Other); University Children's Hospital Basel (Other); Ente Ospedaliero Cantonale, Bellinzona (Other); Kantonsspital Graubünden (Other); University Hospital, Geneva (Other); Centre Hospitalier Universitaire Vaudois (Other); Ostschweizer Kinderspital (Other); Kantonsspital Winterthur KSW (Other); Sanofi (Industry); Hôpital Fribourgeois (Other); University Children's Hospital, Zurich (Other); Luzerner Kantonsspital (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-00377
Record Dates: First submitted 2021-08-04; First posted 2021-08-23 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Optic Neuritis; Transverse Myelitis; Acute Disseminated Encephalomyelitis; Multiple Sclerosis; Neuromyelitis Optica Spectrum Disorder; Anti-NMDAR Encephalitis; Anti-GAD65 Associated Autoimmune Encephalitis; Anti-AMPAR-1/2 Associated Autoimmune Encephalitis; Anti-Lgi-1 Associated Autoimmune Encephalitis; Anti-CASPR-2 Associated Autoimmune Encephalitis; Anti-GABAR-1/2 Associated Autoimmune Encephalitis; Onconeuronal Antibody (Hu, Ri, Yo, Amphiphysin, CRMP-5, Ma-1, Ma-2, SOX-1) Associated Autoimmune Encephalitis; Hashimoto Encephalitis; CNS Vasculitis; CNS Sarcoidosis; CNS Lupus; Rasmussen Encephalitis; Myelin Oligodendrocyte Glycoprotein Antibody-Associated Disease (MOGAD)
MeSH Terms: conditions — Optic Neuritis; Myelitis, Transverse; Encephalomyelitis, Acute Disseminated; Multiple Sclerosis; Neuromyelitis Optica; Anti-N-Methyl-D-Aspartate Receptor Encephalitis; Autoimmune Diseases of the Nervous System; Vasculitis, Central Nervous System; Lupus Vasculitis, Central Nervous System; Encephalitis; Myelin Oligodendrocyte Glycoprotein Antibody-Associated Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 18 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient population: Children, adolescents and adults diagnosed with an IBrainD from 2005 onward and with disease onset before age 18, who are born, treated or living in Switzerland

SUMMARY:
The Swiss-Ped-IBrainD is a national patient registry that collects information on diagnosis, symptoms, treatment, and follow-up of pediatric patients with an inflammatory brain disease in Switzerland. It was first implemented in 2020 in the pediatric clinic of the university hospital in Bern. Further centers all over Switzerland opened for recruitment after that: Aarau, Basel, Bellinzona, Chur, Geneva, Lausanne, Lucerne, St. Gallen, Winterthur and Zurich. The center in Fribourg is expected open for recruitment in 2025. The registry provides data for national and international monitoring and research. It supports research on inflammatory brain diseases in Switzerland and the exchange of knowledge between clinicians, researchers, and therapists. The registry aims to improve the treatment of children with inflammatory brain diseases and optimizing their health care and quality of life.

DETAILED DESCRIPTION:
Background:

Pediatric onset MS and other inflammatory brain diseases (IBrainDs) are severe diseases affecting children and adolescents in a period of essential brain development. This possibly leads to a variety of focal neurological deficits as well as early cognitive impairment. In turn, the cognitive impairment may impact school performance and vocational achievements.

Timely diagnosis and treatment initiation as well as individually tailored management are important for a favorable disease course. However, the diagnosis of the different IBrainDs can be challenging, especially in young children, since their first acute inflammation is often accompanied by unspecific symptoms common to all IBrainDs. A systematic assessment of similarities and differences between clinical signs, symptoms, and diagnostic workup of different IBrainDs will enable faster and more reliable diagnosis.

Furthermore, neither epidemiological data nor information on health care management and disease outcome of pediatric IBrainD patients exist in Switzerland. Therefore, a national registry is being established, which will allow a deeper understanding of pediatric IBrainD epidemiology, clinical presentation, and management. Ultimately, the registry will improve the care of children suffering from an IBrainD in Switzerland.

The Swiss-Ped-IBrainD Registry (title: "Swiss Pediatric Inflammatory Brain Disease Cohort Study", project number: 2019-00377) has been approved by the ethics committees of Bern, the Ethikkommission Nordwest- und Zentralschweiz (EKNZ), the Ethikkommission Ostschweiz (EKOS), and the ethics committees of Zürich, Lausanne, Geneva, and Bellinzona.

Objectives:

The registry pursues the following goals:

1. Gathering representative, population-based epidemiological data on pediatric IBrainD in Switzerland.
2. Monitoring treatment, clinical course, education, social aspects, and outcomes of pediatric IBrainD patients.
3. Providing a platform to facilitate research, national and international collaboration and exchange of knowledge between experts.

The registry thus addresses the increasing requests for medical trial participation and promotes the exchange with existing adult registries (e.g., Swiss MS Registry).

Inclusion/exclusion criteria:

All patients living and/or treated in Switzerland with an IBrainD specified in the following list diagnosed from 2005 onward and with a disease onset before the age of 18.

* Optic neuritis
* Transverse myelitis
* Acute disseminated encephalomyelitis
* Multiple sclerosis
* Neuromyelitis optica spectrum disorders
* Myelin oligodendrocyte glycoprotein antibody-associated disease
* Anti-NMDA-R associated autoimmune encephalitis
* Anti-GAD65 associated autoimmune encephalitis
* Anti-AMPAR-1/2 associated autoimmune encephalitis
* Anti-Lgi-1 associated autoimmune encephalitis
* Anti-CASPR-2 associated autoimmune encephalitis
* Anti-GABAR-1/2 associated autoimmune encephalitis
* Onconeuronal antibody (Hu, Ri, Yo, Amphiphysin, CRMP-5, Ma-1, Ma-2, SOX-1) associated autoimmune encephalitis
* Hashimoto encephalopathy
* CNS vasculitis
* CNS sarcoidosis
* CNS Lupus
* Rasmussen's encephalitis

Excluded are patients with:

1. Neurological symptoms due to infectious diseases of the CNS
2. Genetic/metabolic causes of central demyelinating diseases
3. Neurological symptoms due to Guillain-Barré-Syndrome

Registration of Patients and Collection of Medical Data:

Pediatricians, pediatric neurologists, neurologists, specialists in rehabilitation, and primary care physicians at the participating centers are responsible to identify children with the listed IBrainDs during regular medical consultations. Upon identification, treating physicians inform patients and their parents orally and in writing about the Swiss-Ped-IBrainD. Patients (and their legal representatives if applicable) who want to participate must give their informed consent. Once a patient consents to participate, their medical data will be entered in the registry.

The diagnostic workup and treatment of patients continue as usual and are independent from participation; no examination will be carried out specifically for the Swiss-Ped-IBrainD.

Medical data is collected through the following sources:

* Medical records and reports
* Oral/written information from treating physician
* Oral/written information from patient/family
* Routine statistics and other medical registries
* Questionnaires for patients and families The data collection focuses on diagnostic, follow-up, and relapse variables.

Routine data and linkages:

Communities; Federal Statistical Office (e.g. the birth register, cause of death statistics, hospital statistics)

Current status:

Since 2020, the investigators have included 128 people diagnosed with an IBrainD.

Funding:

* Schweizerische Multiple Sklerose Gesellschaft
* PedNet Bern
* SwissPedRegistry, University of Bern
* Roche Pharma (Switzerland) Ltd
* Novartis Pharma Schweiz AG
* Biogen
* Sanofi
* Anna Mueller Grocholski-Stiftung
* Gottfried und Julia Bangerter-Rhyner Stiftung
* Fondation Johanna Dürmüller-Bol

ELIGIBILITY:
Inclusion Criteria:

All patients living and/or treated in Switzerland with an IBrainD specified in the following list diagnosed from 2005 onward and with a disease onset before the age of 18.

* Written informed consent by patients (and/or legal representative(s), if applicable)
* Optic Neuritis
* Transverse Myelitis
* Acute disseminated encephalomyelitis
* Multiple Sclerosis
* Neuromyelitis Optica Spectrum Disorders
* Myelin oligodendrocyte glycoprotein antibody-associated disease
* Anti-NMDA-R Encephalitis
* Anti-GAD65 Associated Autoimmune Encephalitis
* Anti-AMPAR-1/2 Associated Autoimmune Encephalitis
* Anti-Lgi-1 Associated Autoimmune Encephalitis
* Anti-CASPR-2 Associated Autoimmune Encephalitis
* Anti-GABAR-1/2 Associated Autoimmune Encephalitis
* Onconeuronal Antibody (Hu, Ri, Yo, Amphiphysin, CRMP-5, Ma-1, Ma-2, SOX-1) Associated Autoimmune Encephalitis
* Hashimoto Encephalopathy
* CNS Vasculitis
* CNS Sarcoidosis
* CNS Lupus
* Rasmussen Encephalitis

Exclusion Criteria:

* Neurological symptoms due to infectious diseases of the CNS
* Genetic/metabolic causes of central demyelinating diseases
* Neurological symptoms due to Guillain-Barré-Syndrome

Max Age: 36 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All patients living and/or treated in Switzerland with a listed IBrainD diagnosed from 2005 onward and a disease onset before the age of 18.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-04-14 (Actual); Primary Completion 2071-01-01 (Estimated); Study Completion 2071-01-01 (Estimated)

PRIMARY OUTCOMES:
Personal data | At registration (Life-long; Up to 80 years)
  Registering patient's personal data
Diagnosis | Until reaching of adulthood (0 to 18 years)
  Diagnosis of IBrainD
Age at diagnosis | Until reaching of adulthood (0 to 18 years)
  Age at diagnosis (months and years)
First symptoms | Until reaching of adulthood (0 to 18 years)
  Symptoms before diagnosis
Age at first symptoms | Until reaching of adulthood (0 to 18 years)
  Age at first symptoms
Diagnostic delay | Until reaching of adulthood (0 to 18 years)
  Time elapsed between symptom-onset and diagnosis (days)
Hospitalization | Until reaching of adulthood (0 to 18 years)
  Length of hospitalization at diagnosis or during a relapse (days)
Rehabilitation | Until reaching of adulthood (0 to 18 years)
  Length and type of rehabilitation at diagnosis or during a relapse (days)
Death date | Life-long; Up to 80 years
  Date of death
Death cause | Life-long; Up to 80 years
  Cause of death
Change in EDSS | Until reaching of adulthood (0 to 18 years)
  EDSS change over time
Change in Neurostatus | Until reaching of adulthood (0 to 18 years)
  Neurostatus change over time
Change in medication | Until reaching of adulthood (0 to 18 years)
  Change of IBrainD medication over time
Change in Education | Until reaching of adulthood (0 to 18 years)
  Evolution of education over time
Change in MRI data | Until reaching of adulthood (0 to 18 years)
  Change in number of CNS lesions
Change in MRI data | Until reaching of adulthood (0 to 18 years)
  Change in activity of CNS lesions
Change in laboratory test data | Until reaching of adulthood (0 to 18 years)
  Change in diagnostic markers
Electrophysiological testing | Until reaching of adulthood (0 to 18 years)
  Assessment if the patient did undergo electrophysiological testing.

SECONDARY OUTCOMES:
Future questionnaires | Life-long; Up to 80 years; Will mainly concern childhood (until reaching of adulthood; 0 to 18 years)
  Data from validated instrument such as the Pediatric Quality of Life Inventory (PedsQL); Scale from 0-100, where 100 is the best possible outcome and 0 the worst possible outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Bigi, PD MD, Principal Investigator — ISPM, University of Bern, Bern; Kinderspital Zentralschweiz, Luzern; Sandra Bigi, PD MD, Study Director — ISPM, University of Bern, Bern Kinderspital Zentralschweiz, Luzern
Locations (13):
- Switzerland (13):
  - Kantonsspital Aarau, Aarau, Canton of Aargau
  - Children's Hospital of Eastern Switzerland, Sankt Gallen, Canton of St. Gallen
  - University Children's Hospital Lausanne (CHUV), Lausanne, Canton of Vaud
  - Kantonsspital Winterthur, Winterthur, Canton of Zurich
  - Pediatric Institute of Southern Switzerland, Ospedale San Giovanni, Bellinzona, Canton Ticino
  - Kantonsspital Graubünden, Chur, Kanton Graubünden
  - University Children's Hospital Basel, UKBB, Basel
  - University Children's Hospital, Inselspital Bern, Bern
  - Institute of Social and Preventive Medicine, University of Bern, Bern
  - Hôpital Fribourgeois - Freiburger Spital, Fribourg
  - University Hospitals of Geneva (HUG), Geneva
  - Kinderspital Zentralschweiz, Lucerne
  - University Children's Hospital Zurich, Zurich

IPD SHARING:
Plan to Share IPD: Yes
Researchers who wish to develop a nested study need to submit a proposal to the Swiss-Ped-IBrainD committee and request permission. A concept sheet describing the planned analyses must be approved by the Swiss-Ped-IBrainD committee. Nested studies might need separate ethics permission.

REFERENCES:
- See also: Website of the registry — http://www.swiss-ped-ibraind.ch